CLINICAL TRIAL: NCT01272635
Title: Azithromycin for Preventing the Development of Upper Respiratory Tract Illness Into Lower Respiratory Tract Symptoms in Children and Oral Corticosteroids for Treating Episodes of Significant Lower Respiratory Tract Symptoms in Children
Brief Title: Treatment of Preschool Children With Upper Respiratory Tract Illnesses Using Azythromycin and Lower Respiratory Tract Symptoms Using Oral Corticosteroids.
Acronym: APRIL - OCELOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, dave mauger, Principal Investigator, AsthmaNet Data Coordinating Center, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AsthmaNet 002; 1U10HL098115 (NIH)
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Asthma; Wheezing
Keywords: Asthma; Wheezing; Respiratory Tract Illness; Azythromycin; Prednisolone; Preschool-age
MeSH Terms: conditions — Asthma; Respiratory Sounds | interventions — Azithromycin; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Azythromycin (APRIL) and Prednisolone (OCELOT) (Experimental)
  Interventions: Drug: Azithromycin; Drug: Prednisolone
- Azythromycin (APRIL) and Placebo (OCELOT) (Experimental)
  Interventions: Drug: Azithromycin; Drug: Placebo Prednisolone
- Placebo (APRIL) and Prednisolone (OCELOT) (Experimental)
  Interventions: Drug: Prednisolone; Other: Placebo Azithromycin
- Placebo (APRIL) and Placebo (OCELOT) (Placebo Comparator)
  Interventions: Other: Placebo Azithromycin; Drug: Placebo Prednisolone

INTERVENTIONS:
Drug: Azithromycin — Suspension, 12 mg/kg once daily for 5 days, maximum dose 500mg/day
  Arms: Azythromycin (APRIL) and Placebo (OCELOT); Azythromycin (APRIL) and Prednisolone (OCELOT)
Drug: Prednisolone — Syrup, 1 mg/kg/dose twice daily for 5 days, maximum dose 60mg/day
  Arms: Azythromycin (APRIL) and Prednisolone (OCELOT); Placebo (APRIL) and Prednisolone (OCELOT)
Other: Placebo Azithromycin — Suspension, 12 mg/kg once daily for 5 days, maximum dose 500mg/day
  Arms: Placebo (APRIL) and Placebo (OCELOT); Placebo (APRIL) and Prednisolone (OCELOT)
Drug: Placebo Prednisolone — Syrup, 1 mg/kg/dose twice daily for 5 days, maximum dose 60mg/day
  Arms: Azythromycin (APRIL) and Placebo (OCELOT); Placebo (APRIL) and Placebo (OCELOT)

SUMMARY:
This protocol is comprised of two separate, but linked, clinical trials for treating preschool-aged children with recurrent severe episodes of wheezing. The first study (APRIL) will try to prevent wheezing illness from developing using azithromycin. If a wheezing illness does occur, the second trial (OCELOT) will try to decrease the severity of symptoms using oral corticosteroids.

DETAILED DESCRIPTION:
Preschool aged children often have severe bouts of coughing and/or wheezing that lead to visits to the doctor's office, urgent care, emergency room and often hospitalization. APRIL-OCELOT is a randomized, double-blind, placebo controlled study in 600 preschool children with a history of significant wheezing episodes in the year prior to enrollment. All children enter the APRIL portion of the study, which will compare azithromycin to placebo, given for 5 days during the early signs of an upper respiratory tract illness, for preventing the development of lower respiratory tract symptoms. APRIL is a 78 week study, but participation will end earlier if the child requires a fourth course of APRIL treatment or develops significant lower respiratory tract symptoms. Only those children who develop significant lower respiratory tract symptoms during APRIL will enter the OCELOT portion of the study, which will compare oral corticosteroid to placebo for treating lower respiratory tract symptoms as measured by the Pediatric Respiratory Assessment Measure (PRAM). OCELOT participation will be complete after 14 days. Children may not reenter APRIL after completing OCELOT.

ELIGIBILITY:
Inclusion Criteria:

* 12-71 months of age.
* Recurrent significant wheezing in the past year (any of the following):

  * >3 episodes, ≥1 of which was clinically significant*; OR
  * >2 clinically significant* episodes; OR
  * >4 months of daily controller therapy AND >1 clinically significant* episode.
  * * Clinically significant episode: requiring any of the following: (1) systemic corticosteroids (oral or injectable), (2) unscheduled physician office visit, (3) ED visit, (4) urgent care visit, or (5) hospitalization.
* Up to date with immunizations, including varicella (unless the subject has already had clinical varicella). If the subject needs varicella vaccine, this will be arranged with the primary care physician and must be received prior to randomization.
* Willingness to provide informed consent by the child's parent or guardian.

Exclusion Criteria:

Participants who meet any of the following criteria are NOT eligible for enrollment, but may be re-enrolled if these exclusion criteria are resolved:

* >4 courses of systemic corticosteroids in past 12 months.
* More than 1 hospitalization for wheezing illnesses within the preceding 12 months.
* Use of long-term controller medications for asthma, including inhaled corticosteroids, leukotriene modifiers, cromolyn/nedocromil, or theophylline for more than 8 months (cumulative use) in the past 12 months.
* Current use of higher than step 2 NAEPP asthma guideline therapy (e.g. medium-high dose ICS alone or combination therapy of low-medium-high dose ICS + LABA, montelukast, theophylline or cromolyn). NOTE: children who have evidence of well-controlled symptoms immediately preceding study entry while receiving Step 2 controller therapy (presence of self-reported symptoms on average no more than 2 times per week and less than 2 nights per month of nocturnal awakenings, requiring albuterol, during the 4 weeks preceding visit 1) may be enrolled and will have their controller therapy discontinued upon study entry.
* Use of OCS in the past 2 weeks.
* Daily symptoms or >2 nocturnal awakenings, requiring albuterol, on average in the last 2 weeks.
* Use of antibiotics in the past month.
* Current treatment with antibiotics for diagnosed sinus disease.
* Participation presently or in the past month in another investigational drug trial.
* Evidence that the family may be unreliable or nonadherent, or may move from the clinical center area before trial completion.
* Contraindication of use of systemic corticosteroids or azithromycin.
* Clinically relevant gastroesophageal reflux.
* Concurrent medical conditions other than asthma that are likely to require oral or injectable corticosteroids during the study.
* If receiving allergy shots, change in dose within the past 3 months.

Participants who meet any of the following criteria are NOT eligible for enrollment, and may not be re-enrolled:

* Gestation less than late preterm as defined as birth before 34 weeks gestational age.
* Presence of lung disease other than asthma, such as cystic fibrosis and BPD. Evaluation during the screening process will assure that an adequate evaluation of other lung diseases has been performed.
* Presence of other significant medical illnesses (cardiac, liver, gastrointestinal, endocrine) that would place the study subject at increased risk of participating in the study.
* Immunodeficiency disorders.
* History of respiratory failure requiring mechanical ventilation.
* History of hypoxic seizure.
* History of significant adverse reaction to any study medication ingredient.
* The child has significant developmental delay/failure to thrive, defined as crossing of two major percentile lines during the last year for age and gender. If a child plots less than the 10th percentile for age and gender, a growth chart for the previous year will be obtained from the child's primary care provider.

Ages: 12 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 607 (Actual)
Dates: Start 2011-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Busse, MD, Study Chair — University of Wisconsin, Madison; Leonard B Bacharier, MD, Principal Investigator — Washington University School of Medicine; Fernando D Martinez, MD, Principal Investigator — University of Arizona; David T Mauger, PhD, Principal Investigator — Penn State University; Robert F Lemanske, MD, Principal Investigator — University of Wisconsin, Madison; Wanda Phipatanakul, MD, MS, Principal Investigator — Boston Children's Hospital; Jacqueline Pongracic, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; David Gozal, MD, Principal Investigator — Comer Children's Hospital; James Moy, MD, Principal Investigator — Rush University Medical Center; Stanley Szefler, MD, Principal Investigator — National Jewish Health; Hengameh Raissy, PharmD, Principal Investigator — University of New Mexico; Elizabeth Bade, MD, Principal Investigator — Aurora Sinai Medical Center; Fernando Holguin, MD, Principal Investigator — University of Pittsburgh; James Chmiel, MD, Principal Investigator — Case Western Reserve University School of Medicine; Michael Cabana, MD, MPH, Principal Investigator — University of California, San Francisco; Mindy Benson, PNP, Principal Investigator — UCSF Benioff Children's Hospital Oakland; W. Gerald Teague, MD, Principal Investigator — University of Virginia Health System; Anne Fitzpatrick, MD, Principal Investigator — Emory University
Locations (16):
- United States (16):
  - University of Arizona College of Medicine, Tucson, Arizona
  - Children's Hospital & Research Center Oakland, Oakland, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Center for Urban Population Health, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Fitzpatrick AM, Grunwell JR, Cottrill KA, Mutic AD, Mauger DT. Blood Eosinophils for Prediction of Exacerbation in Preschool Children With Recurrent Wheezing. J Allergy Clin Immunol Pract. 2023 May;11(5):1485-1493.e8. doi: 10.1016/j.jaip.2023.01.037. Epub 2023 Feb 3. PMID 36738927
- [Derived] Bacharier LB, Guilbert TW, Mauger DT, Boehmer S, Beigelman A, Fitzpatrick AM, Jackson DJ, Baxi SN, Benson M, Burnham CD, Cabana M, Castro M, Chmiel JF, Covar R, Daines M, Gaffin JM, Gentile DA, Holguin F, Israel E, Kelly HW, Lazarus SC, Lemanske RF Jr, Ly N, Meade K, Morgan W, Moy J, Olin T, Peters SP, Phipatanakul W, Pongracic JA, Raissy HH, Ross K, Sheehan WJ, Sorkness C, Szefler SJ, Teague WG, Thyne S, Martinez FD. Early Administration of Azithromycin and Prevention of Severe Lower Respiratory Tract Illnesses in Preschool Children With a History of Such Illnesses: A Randomized Clinical Trial. JAMA. 2015 Nov 17;314(19):2034-2044. doi: 10.1001/jama.2015.13896. PMID 26575060

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin/Prednisolone: Active Azithromycin: Suspension, 12 mg/kg once daily for 5 days, maximum dose 500mg/day
  Active Prednisolone: Syrup, 1 mg/kg/dose twice daily for 5 days, maximum dose 60mg/day
- Azithromycin/Placebo: Active Azithromycin: Suspension, 12 mg/kg once daily for 5 days, maximum dose 500mg/day
  Placebo Prednisolone: Syrup, 1 mg/kg/dose twice daily for 5 days, maximum dose 60mg/day
- Placebo/Prednisolone: Placebo Azithromycin: Suspension, 12 mg/kg once daily for 5 days, maximum dose 500mg/day
  Active Prednisolone: Syrup, 1 mg/kg/dose twice daily for 5 days, maximum dose 60mg/day
- Placebo/Placebo: Placebo Azithromycin: Suspension, 12 mg/kg once daily for 5 days, maximum dose 500mg/day
  Placebo Prednisolone: Syrup, 1 mg/kg/dose twice daily for 5 days, maximum dose 60mg/day
Period: Overall Study
Arm/Group | Azithromycin/Prednisolone | Azithromycin/Placebo | Placebo/Prednisolone | Placebo/Placebo
Started | 153 | 154 | 148 | 152
Completed | 122 | 134 | 117 | 129
Not Completed | 31 | 20 | 31 | 23
Not completed — Lost to Follow-up | 31 | 20 | 31 | 23

BASELINE CHARACTERISTICS:
Groups:
- Azythromycin: Azithromycin: Suspension, 12 mg/kg once daily for 5 days, maximum dose 500mg/day
- Placebo: Placebo Azithromycin: Suspension, 12 mg/kg once daily for 5 days, maximum dose 500mg/day
- Total: Total of all reporting groups
Arm/Group | Azythromycin | Placebo | Total
Number analyzed (Participants) | 307 | 300 | 607
Age, Continuous [Mean (Standard Deviation); unit: months] | 41.9 (16.5) | 41.1 (16.4) | 41.5 (16.5)
Gender [Count of Participants; unit: Participants]
  Female | 124 | 118 | 242
  Male | 183 | 182 | 365
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 91 | 92 | 183
  Not Hispanic or Latino | 216 | 208 | 424
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 8
  Asian | 7 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 80 | 77 | 157
  White | 177 | 185 | 362
  More than one race | 40 | 30 | 70
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 307 | 300 | 607
Urgent care or ED visits in prior year [Mean (Standard Deviation); unit: visits] | 2.5 (1.7) | 2.5 (1.6) | 2.5 (1.6)
Wheezing episodes in prior year [Mean (Standard Deviation); unit: episodes] | 4.5 (3.4) | 4.4 (2.9) | 4.5 (3.2)
Hospitalizations for respiratory symptoms in prior year [Median (Inter-Quartile Range); unit: Hospitalizations] | 1 [0 to 4] | 1 [0 to 4] | 1 [0 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Progression to Clinically Significant Lower Respiratory Tract Symptoms
Description: Progression to clinically significant lower respiratory tract symptoms defined by: (1) having symptoms that were more than mild after 3 albuterol administrations over 1 hour, or (2) requiring albuterol administrations more often than once every 4 hours, or (3) requiring more than 6 albuterol treatments over a 24-hour period, or (4) having moderate to severe cough or wheeze for 5 or more days since study medication was initiated.
Time Frame: 14 days after initiation of APRIL therapy
Population: All participants who initiated APRIL therapy
Measure: Number; unit: participants
Arm/Group | Azythromycin | Placebo
Number analyzed (Participants) | 223 | 220
participants | 35 | 57
Statistical Analysis 1: Comparison: Azythromycin vs Placebo; Test type: Superiority or Other; p = 0.04, Discrete time survival analysis; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.41 to 0.98] — Hazard ratio: Numerator is Azithromycin and Denominator is Placebo

2. Primary Outcome: OCELOT: Pediatric Respiratory Assessment Measure
Description: The Pediatric Respiratory Assessment Measure (PRAM) is a composite outcome with scores ranging from 0-12 with higher numbers representing worse symptoms. The score is calculated as the sum total of the follow five elements: (1) scalene retractions, (2) suprasternal retractions, (3) wheezing, (4) air entry, (5) oxygen saturation. A complete description can be found in: Ducharme FM, Chalut D, Plotnick L, et al. The Pediatric Respiratory Assessment Measure: a valid clinical score for assessing acute asthma severity from toddlers to teenagers. J Pediatr 2008;152:476-80.
Time Frame: 36-72 hours after initiation of OCELOT therapy
Population: Participants who developed severe lower respiratory tract infections and initiate blinded OCELOT therapy.
Measure: Mean (Standard Deviation); unit: PRAM score
Groups:
- Prednisone: Active Prednisone: Syrup, 1 mg/kg/dose twice daily for 5 days, maximum dose 60mg/day
- Placebo: Placebo Prednisone: Syrup, 1 mg/kg/dose twice daily for 5 days, maximum dose 60mg/day
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 23 | 21
PRAM score | 0.82 (1.49) | 1.00 (1.41)

3. Secondary Outcome: Asthma Related Symptoms Among RTI Progressing to Severe LRTI
Description: Asthma related symptoms as measured by the parent-completed Pre-school Asthma Symptom Diary (PAD). The PAD was completed daily starting on the first day of an illness and continued until the participant was symptom-free for 2 days. It contains questions of frequency of respiratory symptoms, each scored on a scale of 1 through 7, with higher scores representing increasingly frequent symptoms, with daily scores ranging from 0 (asymptomatic) to a maximum of 102. The total PAD score is the sum of the daily individual symptom scores over the duration of the illness, with higher scores representing more frequent symptoms.
Time Frame: 14 days after initiation of therapy
Population: Respiratory Tract Infections (RTI) progressing to Severe Lower RTI
Measure: Mean (Standard Deviation); unit: PAD score
Arm/Group | Azythromycin | Placebo
Number analyzed (Participants) | 33 | 52
PAD score | 140 (74) | 195 (137)

4. Secondary Outcome: Absence From School, Daycare, and/or Parental Work
Time Frame: 14 days after initiation of therapy
Population: Data were of insufficient quality to be analyzed.
Arm/Group | Azythromycin | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Urgent Care Visits, ED Visits and Hospitalizations
Description: Number of participants who had urgent care visits, ED visits, and/or hospitalizations for respiratory symptoms.
Time Frame: 14 days after initiation of therapy
Population: All participants who initiated APRIL therapy
Measure: Number; unit: participants
Arm/Group | Azythromycin | Placebo
Number analyzed (Participants) | 223 | 220
participants | 20 | 38

6. Secondary Outcome: Drug Related Side Effects
Description: Parent-reported gastrointestinal symptoms during treated RTI.
Time Frame: 14 days after initiation of therapy
Measure: Number; unit: events
Arm/Group | Azythromycin | Placebo
Number analyzed (Participants) | 307 | 300
events | 3 | 1

ADVERSE EVENTS:
Arm/Group | Azythromycin | Placebo
Serious Adverse Events (participants affected / at risk) | 18/307 | 15/300
Other Adverse Events (participants affected / at risk) | 179/307 | 180/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azythromycin (N=307) | Placebo (N=300)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 11 (11)
Acute bronchitis/wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Salmonella (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Viral Enterocolitis (Infections and infestations) | 1 (1) | 0 (0)
Complex Febrile Convulsion (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azythromycin (N=307) | Placebo (N=300)
Acute nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 54 (60) | 43 (47)
Acute Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 75 (93) | 86 (98)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 29 (62) | 30 (59)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (79) | 27 (85)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No